CLINICAL TRIAL: NCT04952532
Title: A Novel Cognitive Remediation Intervention Targeting Poor Decision-Making and Depression in Veterans at High Risk for Suicide: A Safe, Telehealth Approach During the COVID-19 Pandemic
Acronym: CogRemVet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D3738-P; 1I21RX003738-01A1 (NIH)
Record Dates: First submitted 2021-07-02; First posted 2021-07-07 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This is a feasibility and acceptability pilot study which aims to collect preliminary data for a future grant application proposing a randomized clinical trial. This pilot study aims to collect feasibility data of this therapeutic intervention in Veterans. The Neuropsychological Educational Approach to Cognitive Remediation (NEAR, termed CR pus bridging session) intervention involves 20 90-minute sessions (2x/week for 10 weeks). Pre- and post-treatment assessments of neurocognitive, clinical, social, and real-world functioning will be conducted.
Masking Description: This is an open-label pilot study. The clinician conducting the clinical assessments will be blind to how the participants are doing in the treatment intervention. i.e. one clinician will administer the treatment and another will do the outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Remediation+Bridging Intervention (Other): This is a pilot study to collect feasibility data on this novel cognitive remediation intervention for Veterans at high risk for suicide. All patients will receive the active intervention.
  Interventions: Other: Neuropsychological Educational Approach to Cognitive Remediation (NEAR, termed Cognitive Remediation plus Bridging)

INTERVENTIONS:
Other: Neuropsychological Educational Approach to Cognitive Remediation (NEAR, termed Cognitive Remediation plus Bridging) — The proposed study aims to collect pilot data to test the feasibility and acceptability of adjunctive neuroplasticity-based cognitive remediation on key treatment targets. The intervention will be delivered via telehealth to a sample of 36 Veterans with MDD and a history of a suicide attempt. The intervention will be delivered in 20 90-min sessions (2x/week for 10 weeks). Pre-, post, and follow-up assessments will be conducted to assess changes in neurocognitive, clinical, social, and real-world functioning.
  Other Names: Adjunctive Cognitive Remediation

SUMMARY:
Despite large-scale, nationwide efforts to better address suicidal behavior in Veterans at high risk, the development of interventions that target some of the key risk factors associated with suicide remains limited. This study aims to collect pilot data to test feasibility/acceptability of a novel adjunctive evidence-based cognitive remediation (CR) therapy with manualized "Bridging" sessions for transfer and practice of problem-solving strategies for real-world stressors, including those that trigger suicidal thoughts. This 10-week (20 session) Neuropsychological Educational Approach to Cognitive Remediation CR+Bridging telehealth intervention will be administered virtually via HIPPA-compliant services to 36 Veterans with major depressive disorder and a history of suicide attempt(s). Pre-, post-treatment, and follow-up assessments of neurocognitive, clinical, social, and real-world functioning also will be conducted. This study has potential for high public health impact and promise to help improve quality of life for Veterans at high risk for suicide.

DETAILED DESCRIPTION:
Despite large-scale, nationwide efforts to better address suicidal behavior (defined as thoughts and behavior) in high-risk Veterans with major depressive disorder (MDD), the development of interventions that target some of the key risk factors associated with suicide in Veterans with MDD remains limited. That is, while much intervention research continues to investigate treatments like cognitive behavioral therapy (CBT) that target behavioral patterns, emotion processing problems, and cognitive styles associated with suicide risk in MDD, deficits in the neurocognitive substrates that underlie these CBT targets remain under-addressed. Cognitive remediation (CR) and rehabilitation have long been a primary treatment for patients with other psychiatric illnesses, like schizophrenia, for improving cognitive functioning and facilitating transfer of cognitive skills to every-day functioning. However, scant work has examined CR that addresses the neurocognitive deficits underlying suicidal behavior in individuals with MDD. Empirical work has identified key executive functioning (EF) deficits that may be specific to MDD patients with suicidal behavior, and meta-analytic work indicates that CR has moderate effect sizes on cognitive functioning, depression, and daily functioning in MDD. Thus, the field is in dire need of work that examines CR as a recovery-oriented treatment approach for MDD patients at risk for suicide.

The proposed study aims to collect pilot data to test the feasibility and acceptability of adjunctive neuroplasticity-based CR on key treatment targets delivered via telehealth during this time of COVID-19 in a sample of 36 Veterans with MDD and a history of suicide attempt(s). Specifically, it will test the effects of an adjunctive evidence-based cognitive remediation (CR) therapy (adjunctive to treatment as usual) augmented with manualized "Bridging" sessions on transfer and practice of cognitive control and decision-making/problem-solving strategies for real-world situations and problems, including those that trigger suicidal thoughts. The investigators propose to administer the Neuropsychological Educational Approach to Cognitive Remediation (NEAR, termed CR plus "Bridging" session, CR+Bridging) to a total of 36 Veterans with MDD and a history of suicide attempt(s). The intervention will be delivered in 20 90-minute sessions (2x/week for 10 weeks). Pre-treatment assessments of neurocognitive, clinical, social, and real-world functioning will be conducted, including measures that examine the impact of COVID-19 and its accompanying "social-distancing" restrictions. Posttreatment assessments of the same targets will be conducted to determine clinical response to and feasibility of this therapeutic intervention immediately following conclusion of the intervention (Week 10) and at a follow-up assessment (Week 20). This application is novel in that it constitutes the first implementation of this intervention in Veterans with MDD and suicidal behavior. Consistent with RR&D's SPiRE mechanism, this study is high risk, but it has high potential impact and promise to help improve quality of life for Veterans at high risk for suicide.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veteran;
* Primary diagnosis of major depressive disorder (MDD) and a history of suicide attempt in the past year;
* Elevated score (>1SD above the normal mean) on rumination measure (Ruminative Response Scale);
* Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) current suicidal ideation (either passive, i.e. "wish to be dead") or active ideation but with no intent to act on it immediately and no specific plan;
* Currently in psychotherapy treatment as usual (TAU) at the James J. Peters VA Medical Center.
* The investigators will include women and aim for the sample to be 30% women.

Exclusion Criteria:

* Current substance use disorder;
* History of traumatic brain injury; neurological disorder, or other medical confound; compromised intellectual abilities (WASI45 FSIQ<70)
* The investigators will enroll six Veterans in each group and conduct six 10-week intervention cycles for a total sample of 36 Veterans.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin A Hazlett-Oakes, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will request IRB approval to share deidentified data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once the study is completed we will share the supporting information.
Access Criteria: Once the study is completed and data are analyzed and submitted for publication, we will share the deidentified data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Remediation+Bridging Intervention
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Remediation+Bridging Intervention: This is a pilot study to collect feasibility data on this novel cognitive remediation intervention for Veterans at high risk for suicide. All patients will receive the active intervention which is: Active NEAR-S+Bridging intervention.
  Participants were eligible is they were a US Military Veteran and met DSM-5 criteria for a primary psychiatric diagnosis of major depressive disorder based in the SCID-5. More inclusion/exclusion criteria can be found in Goldstein et al 2025; Military Psychology.
Arm/Group | Cognitive Remediation+Bridging Intervention
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 1
  Unknown or Not Reported | 3
Change in Montgomery-Asberg Depression Rating Scale (MADRS) Score: Pre- Minus Post-Tx [Mean (Standard Deviation); unit: Score on a Scale] — A higher MADRS score indicates more severe depression and the overall score ranges from 0 to 60. There are 10 items and each item yields a score of 0 to 6. These 10 sub-items are added together for the total score.
  Score on a Scale | 7.1 (12.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Score: Pre- Minus Post-treatment Intervention
Description: The research team will use the Montgomery-Asberg Depression Rating Scale (MADRS) to examine depression symptoms. A higher MADRS score indicates more severe depression and the overall score ranges from 0 to 60. There are 10 items and each item yields a score of 0 to 6. These 10 sub-items are added together for the total score.
  Typical cutoff points for the total MADRS score are:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20-34 - moderate depression >34 - severe depression Note: The investigators will examine the change in MADRS score from pre-treatment to post-treatment intervention. A positive change score means improvement in depression severity from pre- to post-treatment. The investigators hypothesize that there will be positive change scores following this treatment intervention.
Time Frame: Change in Pre-treatment Score minus Post-treatment Score (Week 10)
Population: Change in pre-treatment MADRS score minus post-treatment score (Week 10)
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- There is Only One Arm in This Acceptability/Feasibility Study and it is the Active Treatment.: Active NEAR-S+Bridging intervention
Arm/Group | There is Only One Arm in This Acceptability/Feasibility Study and it is the Active Treatment.
Number analyzed (Participants) | 9
Score on a Scale | 7.1 (1.6)
Statistical Analysis 1: Comparison: There is Only One Arm in This Acceptability/Feasibility Study and it is the Active Treatment; Test type: Other — Repeated measures ANOVA, F(2,7)=7.6, p<0.05; p < 0.05, ANOVA — This is reported in our peer-reviewed publication: Goldstein et al 2025, Military Psychology

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: We used the same definition of adverse event as clinicaltrials.gov.
Groups:
- Cognitive Remediation+Bridging Intervention: This is a pilot study to collect feasibility data on this novel cognitive remediation intervention for Veterans at high risk for suicide. All patients will receive the active intervention which is: Active NEAR-S+Bridging intervention.
  Participants were eligible is they were a US Military Veteran and met DSM-5 criteria for a primary psychiatric diagnosis of major depressive disorder based in the SCID-5. More inclusion/exclusion criteria can be found in Goldstein et al 2025; Military Psychology.
  There were no adverse events.
Arm/Group | Cognitive Remediation+Bridging Intervention
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
As is the case with pilot studies, results are preliminary due to the study's small sample size and exploratory nature. Thus, the statistical assumptions for repeated-measures ANOVAs may not have been fully met for all analyses. In addition, this pilot study only included male Veterans which may limit generalizability. This study has a small sample size (n=9), which was powered to detect large magnitude effect size improvements (i.e. Hedges' g > 1.0).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT04952532/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04952532/ICF_000.pdf